CLINICAL TRIAL: NCT05773976
Title: An Interventional, Confirmative, Post Marketing Clinical Followup (PMCF) Study to Evaluate Performance and Safety of Ophthalmic Solutions Used to Relieve Dry Eyes Like Symptoms in Glaucoma Patients.
Acronym: M-GLAU-01-2020
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment rate
Sponsor: Montefarmaco OTC SpA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M-GLAU-01-2020
Record Dates: First submitted 2023-02-22; First posted 2023-03-17 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Opthalomology/Dry Eye

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Potential candidates, that according the investigator judgment could be treated with one of IPs (Other): At V0, as per clinical practice, only one of the below reported IPs products can be dispensed to the enrolled subject, depending on investigator clinical evaluation and decision:
  * Afomill Refreshing Soothing
  * Afomill Anti-redness Eye Drops
  * Iridil
  Interventions: Device: Afomill Refreshing Soothing, Afomill Anti-redness Eye Drops, Iridil

INTERVENTIONS:
Device: Afomill Refreshing Soothing, Afomill Anti-redness Eye Drops, Iridil — At baseline visit (V0), as per clinical practice, only one of the below reported IPs products can be dispensed to the enrolled subject, depending on investigator clinical evaluation and decision:
  * Afomill Refreshing Soothing
  * Afomill Anti-redness Eye Drops
  * Iridil

SUMMARY:
Study Rationale: The glaucomas are a group of optic neuropathies characterized by progressive degeneration of retinal ganglion cells. These are central nervous system neurons that have their cell bodies in the inner retina and axons in the optic nerve.

Degeneration of these nerves results in cupping, a characteristic appearance of the optic disc and visual loss. The biological basis of glaucoma is poorly understood and the factors contributing to its progression have not been fully characterized. Glaucoma affects more than 70 million people worldwide with approximately 10% being bilaterally blind, making it the leading cause of irreversible blindness in the world. Glaucoma can remain asymptomatic until it is severe, resulting in a high likelihood that the number of affected individuals is much higher than the number known to have it.

The tear film is fundamental in the maintenance of the ocular surface. Any condition that adversely affects the stability and function of the tear film such as dry eye symptom, blepharitis, and meibomian gland dysfunction, dysfunctional tear film syndrome, or toxicity of topical medications may result in onset of an ocular surface disease (OSD). The symptoms of OSD may include dryness, burning or stinging, itching, irritation, tearing, photophobia, foreign-body sensation, grittiness, redness, fatigue, fluctuating visual acuity, and blurred vision.

OSD is a common comorbidity in glaucoma patients in part due to the fact thatits prevalence as in glaucoma increases with age. OSD is seen in approximately 15% of the general elderly population and is reported in 48% to 59% of patients with medically treated glaucoma. One in six patients with glaucoma has OSD symptoms severe enough that they need some form of treatment.

Ophthalmic solutions with soothing and refreshing proprieties, as addon treatment to glaucoma therapy, could relieve the OSD symptomatology, dry eye like, in glaucoma patients, improving their quality of life.

For these reasons, an interventional, confirmative, post marketing clinical followup (PMCF) study was planned to evaluate the performance and safety of ophthalmic solutions used to relieve dry eyes like symptoms in glaucoma patients.

Study Objective: The objectives of this PMCF study are confirmation of the performance, collection of additional safety data regarding expected adverse events and detection of potential unexpected adverse events associated with use of three investigational products (IPs).

The IPs are on the market with the following brand names:

* Afomill Refreshing Soothing
* Afomill Anti-redness Eye Drops
* Iridil

DETAILED DESCRIPTION:
Study Rationale: The glaucomas are a group of optic neuropathies characterized by progressive degeneration of retinal ganglion cells. These are central nervous system neurons that have their cell bodies in the inner retina and axons in the optic nerve.

Degeneration of these nerves results in cupping, a characteristic appearance of the optic disc and visual loss. The biological basis of glaucoma is poorly understood and the factors contributing to its progression have not been fully characterized. Glaucoma affects more than 70 million people worldwide with approximately 10% being bilaterally blind, making it the leading cause of irreversible blindness in the world. Glaucoma can remain asymptomatic until it is severe, resulting in a high likelihood that the number of affected individuals is much higher than the number known to have it.

The tear film is fundamental in the maintenance of the ocular surface. Any condition that adversely affects the stability and function of the tear film such as dry eye symptom, blepharitis, and meibomian gland dysfunction, dysfunctional tear film syndrome, or toxicity of topical medications may result in onset of an ocular surface disease (OSD). The symptoms of OSD may include dryness, burning or stinging, itching, irritation, tearing, photophobia, foreign-body sensation, grittiness, redness, fatigue, fluctuating visual acuity, and blurred vision.

OSD is a common comorbidity in glaucoma patients in part due to the fact thatits prevalence as in glaucoma increases with age. OSD is seen in approximately 15% of the general elderly population and is reported in 48% to 59% of patients with medically treated glaucoma. One in six patients with glaucoma has OSD symptoms severe enough that they need some form of treatment.

Ophthalmic solutions with soothing and refreshing proprieties, as addon treatment to glaucoma therapy, could relieve the OSD symptomatology, dry eye like, in glaucoma patients, improving their quality of life.

For these reasons, an interventional, confirmative, post marketing clinical followup (PMCF) study was planned to evaluate the performance and safety of ophthalmic solutions used to relieve dry eyes like symptoms in glaucoma patients.

Study Objective: The objectives of this PMCF study are confirmation of the performance, collection of additional safety data regarding expected adverse events and detection of potential unexpected adverse events associated with use of three investigational products (IPs).

The IPs are on the market with the following brand names:

* Afomill Refreshing Soothing
* Afomill Anti-redness Eye Drops
* Iridil

Primary • To evaluate the performance of IPs used as intended to relieve dry eye like symptoms in glaucoma patients.

Secondary

* To evaluate the performance of IPs used to affect the tear film in glaucoma patients.
* To evaluate the efficacy of IPs used as intended to relieve symptoms of OSD in glaucoma patients.
* To evaluate the maintenance of the basic condition of intraocular pressure in glaucoma patients.
* To evaluate the safety and tolerability of the IPs.
* To evaluate the patient satisfaction of the IPs.

Methodology: Potential candidates, that according the investigator judgment could be treated with one of IPs, will be identified, with the assessment of their eligibility criteria. Each subject, after signing the Informed Consent Form, will enter the screening and baseline phase (the 2 visits will coincide) during which baseline procedures will be completed.

At baseline visit (V0), as per clinical practice, only one of the below reported IPs products can be dispensed to the enrolled subject, depending on investigator clinical evaluation and decision:

* Afomill Refreshing Soothing
* Afomill Anti-redness Eye Drops
* Iridil

The patient will perform 2 on site visits: V0 and V2/EOS. To monitor the safety, 1 phone contact is planned (V1) to check for potential adverse events and concomitant medications intake.

Data coming from additional assessments (e.g. blood tests), if done per clinical practice to perform glaucoma diagnosis and evaluations, might be collected and used.

Planned: About 90 patients in total.

Treatment duration: After baseline visit and IP dispensing, the treatment duration (according to the Investigation Product IFU) will be prolonged until the V2 (EOS visit; 30+ 5 days).

The "Safety Analysis Set" (SAS): this set included all enrolled patients who took at least one dose of IP.

The "Full Analysis Set" (FAS): this set included all enrolled patients who took at least one dose of IP, and with a baseline and at least one post-baseline performance assessment.

The "Per-Protocol" (PP) set: would include all the FAS patients who (a) met all inclusion/exclusion criteria liable to affect the performance assessment, (b) did not present serious deviations of the protocol that may affect efficacy.

Dose/dosage: All IPs are available as preservative-free 0,5 ml single-dose vials.

Afomill Refreshing Soothing and Afomill Anti-redness Eye Drops are also available as preservative free 10 ml multi-dose bottle.

Iridil is also available as 10 ml multi-dose bottle containing vanishing preservative (sodium chlorite).

The IP dosage for each individual case will be defined according to investigator judgment.

Administration: The application of IP on eye surface should be performed in accordance to the indication for use. The use of IP will be an add-on therapy to the glaucoma treatment prescribed as per clinical practice. According to the Investigator judgement, based on the subject clinical conditions and the indications reported on the IFU of IPs, one of the investigational products can be dispensed to the subject to be enrolled in the trial. The first administration and the intervals at which the treatment should be repeated, to be done as per investigator judgment and according the IFU, depend on various factors regarding the physiology of the patients (e.g. type of eye-tear film, anatomy, age), their lifestyle (e.g. use of computer, wearing of contact lenses).

Primary efficacy endpoint

• To evaluate the performance of IPs to relieve symptoms of OSD (dry eye like symptoms, e.g. burning, redness, fatigue, or irritation sensation according the IFU) in glaucoma patients, the Shirmer I test (ST) might be completed at baseline (V0) and end of study visit (EOS/V2). The evaluation will be performed stratified by study IPs.

Secondary efficacy endpoints

* To evaluate the performance of IPs to affect the tear film in glaucoma patients, the Tear breakup time (TBUT) test might be completed at baseline (V0) and end of study visit (EOS/V2). The evaluation will be performed stratified by study IPs.
* To assess the efficacy of IPs used as intended to relieve symptoms of OSD (dry eye like symptoms, e.g. burning, redness, fatigue, or irritation sensation according the IFU) in glaucoma patients, the difference of "Ocular surface index" (OSDI) Questionnaire between baseline (V0) and end of study visit (EOS/V2) will be evaluated stratified by study IPs.
* The maintenance of the basic condition of glaucoma will be evaluated with Intraocular pressure (IOP) values
* To evaluate the safety and tolerability of the IPs a Visual Analogue Scale (VAS) will be used.
* The patient satisfaction will be evaluated with a 5-points Likert Scale.

Safety will be monitored through eye examination and adverse events including assessment of relationship to the IP.

Time-points for efficacy and safety: Baseline (V0) and follow up visit(s) performed.

Statistical methods: Supposing a minimum difference of 10% between after treatment and at baseline visit in terms of mean ST value, with a standard deviation (SD) equal to 3 mm/5 min, a correlation between baseline and end of treatment of 80%, and a type I error of 5%, 25 patients are sufficient to reach a statistical power greater than 80% for each IPs.

Moreover, planning to enroll a total of 30 patients would allow for a 15% dropout rate. Considering all IPs included, 90 patients should be enrolled in the study.

In general, all the variables will be descriptively analyzed by treatment groups and visit (mean, median, standard deviation, minimum and maximum for continuous variables after normality check of distribution with Kolmogorov- Smirnov test, frequency distribution for categorical variables). All the analysis will be detailed in the Statistical Analysis Plan (SAP) which will be finalized in Version 1.0 before the Data Base Lock (DBL).

In details, the safety data will include (at least) physical examinations, laboratory data and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patient Informed consent form (ICF) signed;
* M & F Aged ≥ 18 years at the time of the signature of ICF;
* Patients with a prescription, as per clinical practice, of a topic treatment for glaucoma or ocular hypertension (i.e. anti-hypertensive eye drops), showing OSD symptoms (dry eye like symptoms; e.g. burning, redness, fatigue, or irritation sensation).
* Willing not to use other eye drops during the entire treatment period (except for the possible drug-containing glaucoma treatment prescribed as per clinical practice).

Exclusion Criteria:

* Other - different - eyes clinical conditions;
* Retinal pathology;
* Other type of ophthalmic neuropathy;
* Severe POAG;
* Known hypersensitivity or allergy to IP components;
* Eye surgery during the previous 6 months (e.g. cataract surgery)
* Presence of any relevant severe organic, systemic or metabolic disease (particularly significant history of cardiac, renal, neurological, psychiatric, oncology, endocrinology, metabolic or hepatic disease), or abnormal laboratory values that will be deemed clinically significant in Investigator's opinion;
* Participation in another investigational study;
* Inability to follow all study procedures, including attending all site visits, tests and examinations;
* Mental incapacity that precludes adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Evaluate the performance of Investigational Products to relieve symptoms of ocular surface disease in glaucoma patients. The performance will be evaluated by Shirmer I test at baseline (V0) and end of study visit (change will be assessed) | Day 0 (baseline visit the IP will be dispensed) and Day 30
  To evaluate the performance of IPs to relieve symptoms of OSD (dry eye like symptoms, e.g. burning, redness, fatigue, or irritation sensation according the IFU) in glaucoma patients, the Shirmer I test (ST) might be completed at baseline (V0) and end of study visit (EOS/V2). The evaluation will be performed stratified by study IPs.

SECONDARY OUTCOMES:
Evaluate the performance of Investigational Products to affect the tear film in glaucoma patients. The performance will be evaluated by Tear breakup time test at baseline (V0) and end of study visit (change will be assessed) | Day 0 (baseline visit the IP will be dispensed) and Day 30
  To evaluate the performance of IPs to affect the tear film in glaucoma patients, the Tear breakup time (TBUT) test might be completed at baseline (V0) and end of study visit (EOS/V2). The evaluation will be performed stratified by study IPs.
Efficacy of Investigational Products used as intended to relieve symptoms of OSD in glaucoma patients. The Efficacy will be evaluated by Questionnaire at baseline (V0) and end of study visit (change will be assessed) | Day 0 (baseline visit the IP will be dispensed) and Day 30
  To assess the efficacy of IPs used as intended to relieve symptoms of OSD (dry eye like symptoms, e.g. burning, redness, fatigue, or irritation sensation according the IFU) in glaucoma patients, the difference of "Ocular surface index" (OSDI) Questionnaire between baseline (V0) and end of study visit (EOS/V2) will be evaluated stratified by study IPs.
Evaluation of the maintenance of the basic condition of glaucoma by Intraocular pressure at baseline (V0) and end of study visit (change will be assessed) | Day 0 (baseline visit the IP will be dispensed) and Day 30
  The maintenance of the basic condition of glaucoma will be evaluated with Intraocular pressure (IOP) values
To evaluate the safety and tolerability of the Investigational Products by Visual Analogue Scale at the end of study visit | Day 30
  To evaluate the safety and tolerability of the IPs a Visual Analogue Scale (VAS) will be used.
The patient satisfaction will be evaluated with a 5-points Likert Scale at the end of study visit | Day 30
  The patient satisfaction will be evaluated with a 5-points Likert Scale.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Istituto Auxologico Italiano, Milan
  - Ospedale Felice Liotti Pontedera, Pisa